CLINICAL TRIAL: NCT05191316
Title: the Efficacy and Safety of th 3-steps Conservative Approach in the Management of Placenta Accreta Spectrum (a Novel Technique)
Brief Title: the Efficacy and Safety of the 3-steps Conservative Approach in the Management of Placenta Accreta Spectrum (a Novel Technique)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Essameldin Mohamed Abdullah, DR., Cairo University
Other Study IDs: MEMAbdullah
Record Dates: First submitted 2021-12-12; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Placenta Accreta, Third Trimester
Keywords: surgical conservative management
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Placenta accrete spectrum (PAS) is an heterogeneous condition associated with a high maternal morbidity and mortality rate, presenting unique challenges in its diagnosis and management (Morlandoi et al., 2020). PAS describes a clinical situation where the placenta does not detach spontaneously after delivery and cannot be forcibly removed without causing massive and potentially life-threatening bleeding (Jauniaux et al., 2018), in this study we study a novel 3-step technique for surgical conservative management of PAS, in terms of efficacy and safety.

DETAILED DESCRIPTION:
* Informed written consent: after discussing the nature of the study as well as the expected value, outcome, and possible adverse effects.
* Full medical history: including full obstetric history and current pregnancy history (entailing the 1st day of LMP).
* Thorough Clinical Examination: general (maternal body weight and vital signs) and full obstetric examination.
* Obstetric ultrasonography: to confirm gestational age and the eligibility of the current pregnancy to participate in the study together with full placental assessment (diagnosis of PAS - placentation site and vasculature - extent of invasion to myometrial wall and surrounding structures as bladder wall invasion), with intra-operative confirmation aided by whether placental separation will occur or not.
* Preoperative laboratory tests: including prothrombin time, prothrombin concentration, complete blood count, and liver and kidney function tests.
* Operative steps: (A novel conservative 3 step technique)

  * Patient positioning: under spinal anesthesia, the patient will be placed in the dorsal supine position. The patient will be then prepped and draped in the usual fashion for an abdominal procedure.
  * A vertical midline incision will be done.
  * Abdominal wall will be dissected in layers using sharp dissection or electro-coagulation instruments till the entry of peritoneal cavity.
  * Dissection and release of the adherent bladder from the anterior uterine wall as low as possible (vesico-uterine peritoneal fold) together with the vascular disconnection of the newly formed vessels connecting the adherent invasive placenta to the urinary bladder. Dissection will be carried out laterally until both ureters are reached out and identified and in the midline until the lower edge of the placenta is identified.
  * Transverse uterine incision above the upper border of placenta will be done followed by delivery of the fetus and immediate cord clamping (< 30 seconds) then the uterus will be exteriorized without trying to separate the adherent placenta and the uterine incision will be approximated by four towel clips (to reduce the blood loss).
  * Placental bed devascularization (step 1): ligation of uterine arteries on two levels (one immediately under the lower level of placenta and another at least 5 mm above the upper edge of the adherent part of the placenta (superior-vesical arteries, feeding vessels of the placenta invading the back of the bladder will be also ligated).
  * Cervical control sutures (step 2): transverse suture (full thickness) in the lower uterine segment at least 5 mm below the lower border of the placenta with or without similar stitch in the posterior uterine wall just above the uterosacral ligaments attachments.
  * Delivery of the placenta with trimming of the invaded parts of the myometrium (step 3) followed by compression sutures taken in bleeding placental bed (if present) then myometrial reconstruction is done via continuous suture and mattress sutures.
  * Bilateral ligation of the internal iliac arteries (4 cm distal to its origin) will be done if there is insufficient hemostasis is still present in spite of the above-mentioned steps to enhance further pelvic devascularization or if there's frank bladder invasion.
  * In case of uncontrolled bleeding or failed the above-mentioned measures, hysterectomy will be done.
  * Closure of abdominal wall in layers
* For all patients, 1 gm (10 ml) Tranexamic acid (Kapron, Amoun, Egypt) diluted in 20 ml of Glucose 5% will be given as intravenous infusion over 5 minutes, at least 15 minutes prior to skin incision in addition to 400 microgram misoprostol (2 tablets - Cytotec, Pfizer, G.D. Searle LLC) will administered rectally together with catheter insertion. Following the delivery of the baby, patients will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500mL lactated Ringer's solution (infused at a rate of 125mL/h).
* The operative steps (operative procedure, operative time, time interval between skin incision and fetal delivery, internal iliac artery ligation) will be recorded. The number and the difference of weight of operative towels (before and after CS) and amount of blood in suction unit will be also recorded.
* The received blood units or blood products will be recorded (intra or postoperative).
* Fluid monitoring will be performed through rate of infusion and urine output.
* The neonatal outcome (APGAR at 1 and 5 minutes, NICU admission and neonatal death) will be recorded.
* A complete blood count will be performed 12 hours after delivery. All patients will be followed up following the delivery as regard occurrence of primary postpartum hemorrhage (within the first 24 hours), re-exploration with further surgical procedures, the need for additional blood transfusion (within the first 24 hours) or ICU admission.
* Estimated Blood Loss (EBL) was evaluated as follows:

A. The number of operative towels used. B. The difference of weight of operative towels (before and after CS) plus the amount of blood in suction unit (we calculated 1 gram of weight difference equal to 1 ml blood loss).

C. EBL calculation according to the following formula:

EBL= EBV x Preoperative hematocrit- Postoperative hematocrit Postoperative hematocrit Where EBV is estimated blood volume of the patient in mL (equals weight in kg × 85).

* At least 6 weeks post-operatively, a 2D and 3D ultrasonographic assessment of the uterus will be done, assessing the uterine cavity (the presence and extend of a uterine niche). Trans-abdominal ultrasound complimented with trans-vaginal ultrasound, by an expert, using a Voluson E8 Expert (GE Healthcare Ultrasound Korea, Ltd) ultrasound will be done. All ultrasound findings will be recorded.
* Patients who the 3-step management fail and are managed by a cesarean hysterectomy will be considered and recorded as failed and will be excluded from the study.
* In avoidance of false positive PAS, an intra-operative confirmation will be done, should full placental separation or complete placenta accrete be found, those patients will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-40 years old.
* Pregnant females with previous CS deliveries (at least 1) diagnosed with focal or partial PAS (placenta accreta/increta/percreta) candidate for 3rd trimester cesarean delivery.
* Patients wishing uterine conservation to preserve fertility.
* Gestational age: > 28 weeks confirmed by the 1st day of the LMP or 1st trimesteric ultrasound scan.
* Singleton pregnancies.
* CS under general anesthesia.

Exclusion Criteria:

* Maternal Anemia (hemoglobin < 10 g %).
* Chronic or pregnancy induced medical disorders (e.g., cardiac, renal, DM and hepatic diseases).
* Patients presented with severe antepartum hemorrhage.
* Patients requested radical management (caesarean hysterectomy).
* Fetal death (IUFD).
* Fetal anomalies or IUGR (estimated fetal weight below the 5th centile).
* Women attending for emergency CS.
* Patients found to be suffering from placenta previa or total placenta accreta

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 28 pregnant females diagnosed with focal or partial PAS (placenta accreta/increta/percreta) undergoing 3rd trimester cesarean delivery.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the 3-steps conservative approach as a novel technique in the management of PAS (measured using the percentage of successful surgical procedure among study population). | 6 weeks
  immediate and short term success of the 3-step conservative management technique

SECONDARY OUTCOMES:
estimated blood loss (EBL) | pre and post operative
  To evaluate the rate and amount of blood and blood product transfusion
evaluate the rate of complication | first 24 hrs post operative
  primary postpartum hemorrhage, re-exploration with further surgical procedures, the need for additional blood transfusio or ICU admission.
To evaluate the impact of the studied approach on the integrity of uterine cavity | 6 weeks post-operative
  (the presence of niche) follow up CS scar US examination for the presence of a uterine niche, which may affect future pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Gaafar, M.D, Principal Investigator — prof. of obstetrics and gynecology (Faculty of medicine -Cairo university); Moataz M El-sherbini, M.D, Principal Investigator — prof. of obstetrics and gynecology (Faculty of medicine -Cairo university); Abdalla m Mousa, M.D, Principal Investigator — lecturer of obstetrics and gynecology (Faculty of medicine -Cairo university); mostafa E Abdalla, MRCOG, Principal Investigator — Senior specialist clinical fellow, gynecology Guy's and St. Thomas's NHS TRUST; Mazen m Abdel-rasheed, PhD, Principal Investigator — reproductive health research department, national research centre; sondos m salem, PhD, Principal Investigator — reproductive health research department, national research centre
Locations (1):
- Kasr al Ainy university, obstetrics and gynecology department, Cairo, Greater-cairo, Egypt